CLINICAL TRIAL: NCT05999734
Title: Ultrasound-Guided Mid-Transverse Process to Pleura Block for Analgesia in Pediatric Thoracotomy: A Randomized Controlled Study
Brief Title: Mid-transverse Process to Pleura Block in Pediatric Thoracotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Salah Eldin Gawish, Principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTP block
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Ultrasound Guided Block; Pediatric Surgery; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing pediatric thoracotomy will receive general anesthesia alone. (No Intervention): the patients will receive general anesthesia alone. Anesthesia will be induced by inhalation of sevoflurane at 8% concentration which will decreased gradually down to 2% concentration carried by 100% oxygen, with loss of consciousness; a peripheral intra venous cannula with suitable size will be inserted, then the neuromuscular blockade will be facilitated by cisatracurium 0.15 mg/ kg to allow tracheal intubation with appropriate sized endotracheal tube. Fentanyl 1μg/ kg will be given and anesthesia will be maintained with air and O2 (50:50) and along with 2% end tidal concentration of sevoflurane to control the depth of anesthesia. At the end of surgery residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and extubation will be performed after complete recovery of the airway reflexes.
- general anesthesia and ultrasound guided MTP block (Active Comparator): midpoint between the transverse process and the pleura 0.5mL/kg 0.25% bupivacaine will be injected.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Before skin incision, under complete aseptic precautions and sterilization, the patient will be placed in a lateral position. The spinous process of the fourth thoracic vertebra will be identified and marked. The ultrasound guided MTP block will be done by high frequency linear transducer will be placed in position just lateral to the spinous processes of thoracic vertebra target of the paravertebral space. A 50 mm 22-gauge echogenic needle will be inserted in an in plane technique from a caudal to a cephalad direction and will be advanced. When the needle tip reaches the midpoint between the transverse process and the pleura, 1 ml normal saline will be injected. Once the needle tip has been confirmed and after careful aspiration to demonstrate the absence of air or blood, 0.5mL/kg 0.25% bupivacaine will be injected.
  Other Names: Mid transverse process to pleural block
  Arms: general anesthesia and ultrasound guided MTP block

SUMMARY:
The aim of this study is to assess the effectiveness of analgesia of US guided MTP block in pediatrics undergoing thoracotomy.

DETAILED DESCRIPTION:
Pain following surgery is a universal phenomenon which up to now is often underestimated and undertreated especially in pediatrics. Any postoperative analgesic technique should meet three criteria, which are effectiveness, universal applicability and safety.

Thoracotomy is widely known to cause severe acute pain. This pain can be very distressing for both children and their parents. If not treated properly, it may acutely cause ventilation-perfusion disorder and hypoxemia, together with a change in lung mechanics. It may lead to a delay in recovery, with some long-term sequelae. As a part of multimodal analgesia, many regional blocks have been described.

Regional anesthesia techniques are increasingly used in all surgical settings. Even in the context of thoracic surgery, new peripheral regional anesthesia techniques are being tested as alternatives to those already used. This proliferation of new techniques is explained, on the one hand, by the evolution of surgical techniques, which are becoming less and less invasive, and on the other hand, by the frequency and severity of the complications induced by thoracic epidural anesthesia and paravertebral block - currently the gold standards in context of pediatric setting.

Paravertebral block (PVB) has gained more popularity than other regional analgesic techniques including epidural for perioperative analgesia in pediatric surgery. Thoracic PVB provides adequate postoperative analgesia with favorable adverse effects. The use of thoracic PVB is associated with decreased pain severity and opioid consumption in both adults and children.

Many clinicians hesitate to apply the PVB technique due to the risk of serious complications such as pneumothorax. Therefore, the safest and most effective methods are being tried by clinicians. In a study conducted on cadavers claimed that mid-transverse process to pleura (MTP) block (an injection point midway between the pleura and posterior border of the transverse process) provides a paravertebral block due to the paravertebral spread of the local anesthetic agent through fenestrations and septations in the superior costotransverse ligament. They thought that MTP block may be as effective as PVB in postoperative pain management with less risk of possible complications.

ELIGIBILITY:
Inclusion Criteria:

* The study will include 50 pediatric patients of both sexes aged from 5 to 15 years old with American Society of Anesthesiologists physical status I& II undergoing elective open thoracotomy.

Exclusion Criteria:

* Refusal of parents.
* Repeated thoracotomy.
* Emergency surgery.
* Mechanically ventilated patients.
* Bleeding disorders.
* Allergy to study drugs.
* Infection at the site of the needle puncture.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The total dose of morphine consumption in the first postoperative 24 hours. | 24 hours postoperative
  The total dose of morphine consumption in the first postoperative 24 hours.

SECONDARY OUTCOMES:
Pain will be assessed by the face, legs, activity, cry and consolability (FLACC) score in children at 1, 2, 6, 12, 18 and 24 hours postoperative. | 1, 2, 6, 12, 18 and 24 hours postoperative.
  Pain will be assessed by the face, legs, activity, cry and consolability (FLACC) score in children at 1, 2, 6, 12, 18 and 24 hours postoperative.The scale is scored in a range of 0 to 10 with 0 representing no pain, 10 representing the maxim
Total intraoperative fentanyl consumption (μ/kg) starting from induction of anesthesia till the end of surgery. | from induction of anesthesia till the end of surgery.
  Total intraoperative fentanyl consumption (μ/kg) starting from induction of anesthesia till the end of surgery.
Diaphragmatic excursion will be measured preoperative and postoperative in post anesthesia care unit (PACU). | Immediately 15 minutes preoperative and 15 minutes postoperative
  Diaphragmatic excursion will be measured preoperative and postoperative in post anesthesia care unit (PACU).

IPD SHARING:
Plan to Share IPD: No